CLINICAL TRIAL: NCT04419324
Title: A Pilot Study to Evaluate the Use of a Transoral Flexible Endoscope With Magnifying Narrow Band Imaging in Nasopharyngeal Cancer
Brief Title: To Evaluate Transoral Flexible Endoscope With Narrow Band Imaging in Nasopharyngeal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jason Chan, Prof. Chan, Jason Ying Kuen, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 01
Record Dates: First submitted 2020-05-31; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: This is a case-control pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- esophago-gastroscopy endoscopy with narrow band imaging (Other): a transoral flexible endoscope with magnifying narrow band imaging in nasopharyngeal examination
  Interventions: Device: transoral flexible endoscope with magnifying narrow band imaging

INTERVENTIONS:
Device: transoral flexible endoscope with magnifying narrow band imaging — To use an esophago-gastroscopy endoscope (OGD) with Narrow Band Imaging (NBI) passed transorally and retroflexed into the nasopharynx to view the nasopharynx with increased magnification and clarity for the diagnosis of nasopharyngeal carcinoma.

SUMMARY:
Nasopharyngeal carcinoma (NPC) is endemic in our region and is the 9th most common cancer in Hong Kong. Traditionally diagnosis has been through a nasoendoscopic examination of the nasopharynx with white light followed by a biopsy of suspicious lesions for a confirmatory diagnosis. However, given the geometry of the anatomy of the nasopharynx, with its inherent crevices and varying amounts of lymphoid tissues, lesions are not always easily identified leading to potential missed lesions. The non-specific aspect of white light also leads to excessive biopsies that are not without risk and of some discomfort to patients. Recent advances in liquid biopsies have also allowed for the detection of earlier and smaller lesions that are not always easily identified on nasoendoscopy but rather are seen on Magnetic Resonance Imaging (MRI)1 .

An alternative imaging technique is the use of Narrow Band Imaging (NBI) to view the vasculature of the mucosa to identify suspicious lesions for pre-malignancy and malignancy that has been popularized in the gastrointestinal tract. In NPC, NBI with the flexible nasoendoscopes has been used in the diagnosis of NPC with varying success2-5 . Our own group's research has found that in NPC NBI has limitations arising from a lack of consensus on vascular findings on NBI that constitute malignancy, lack of magnification and long focal length of current nasoendoscopes5-8 . Flexible endoscopy using conventional esophago-gastroscopy endoscope (OGD) with NBI and magnification power up to 80x overcome the limitations of current nasoendoscopes, however their size precludes the passing of these endoscopes through the nasal cavity.

Here in this pilot study we will seek to use an OGD with NBI passed transorally and retroflexed into the nasopharynx to view the nasopharynx with increased magnification and clarity to evaluate the feasibility of this study in the diagnosis of nasopharyngeal carcinoma.

Study questions:

1. Is it feasible to use an OGD with magnifying NBI for the diagnosis of NPC?
2. Are there features detected on NBI OGD that are diagnostic of NPC?
3. Do histological features correspond with NBI findings?

DETAILED DESCRIPTION:
This is a case-control pilot study. We will recruit 40 patients. 20 patients with newly diagnosed primary NPC will be recruited to the test group. 20 patients undergoing an OGD for lesions not involving disease of the head and neck region will be recruited to the control group.

NBI OGD and flexible nasoendoscopy will be performed to examine patients' nasopharyngeal region.

NBI OGD: Endoscopic procedures would be performed by our investigators with expertise on performing upper endoscopy. Endoscopes with magnification and NBI function would be used (GF-H290Z, Olympus Medical Corporations, Tokyo, Japan). A soft black hood would be attached to the tip of the endoscope for better focal length adjustment.

Upon insertion through a mouthpiece, the scope will then be retroflexed into the nasopharynx and the lateral walls into the Fossa of Rosenmuller and the posterior nasopharyngeal wall will be systematically examined with white light and NBI. Target suspicious areas would be examined by use of magnification with the power up to 80X.

Flexible nasoendoscopy: The nasoendoscope is introduced into the nose, the nasal cavity and nasopharyngnx. It has a camera and a light at the end and allows our doctor to check for any abnormal looking areas. Upon identification of suspicious lesion. Biopsies of sites with different NBI findings will be taken to correlate the NBI findings with histological features.

ELIGIBILITY:
General Inclusion Criteria for both study groups, Test group and Control group.

1. No previous radiotherapy to the head and neck region
2. 18 Years and older
3. Able to provide informed consent
4. No cognitive impairment

Test group - Specific Inclusion Criteria 1) Newly diagnosed primary nasopharyngeal carcinoma

Control group - Specific Inclusion Criteria

1) Patients undergoing an OGD for lesions not involving disease of the head and neck region

General Exclusion Criteria for both study groups, Test group and Control group.

1. On anticoagulation including Plavix, warfarin and NOAC's
2. Current mucosal lesions of the head and neck region
3. History of malignancy
4. Concomitant malignant disease
5. Trismus preventing an OGD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The vasculature of the nasopharyngeal region | during enrollment period
  The vasculature of the nasopharyngeal region which capture by the transoral flexible endoscope with magnifying narrow band imaging

SECONDARY OUTCOMES:
Histological features of nasopharyngeal lesion | during enrollment period
  Histological features of nasopharyngeal biopsy which is done during endoscopy with magnifying narrow band imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chan, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No